CLINICAL TRIAL: NCT00742729
Title: Increasing Colorectal Cancer Screening Among Filipino Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: American Cancer Society, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: RSGT-04-210-01-CPPB
Record Dates: First submitted 2008-08-27; First posted 2008-08-28 (Estimated); Last update posted 2016-08-01 (Estimated); Status verified 2010-11

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening; Fecal occult blood test; Endoscopies; Filipino American immigrants; Community based organizations and churches
MeSH Terms: conditions — Colorectal Neoplasms | interventions — DMAC2L protein, human

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental): Educational small group session with free FOBT kit
  Interventions: Behavioral: Arm 1
- Arm 2 (Experimental): Educational small group session with no FOBT kit
  Interventions: Behavioral: Arm 2
- Arm 3 (Sham Comparator): Control
  Interventions: Behavioral: Arm 3

INTERVENTIONS:
Behavioral: Arm 1 — Educational small group session with free FOBT kit
  Other Names: Intervention 1
  Arms: Arm 1
Behavioral: Arm 2 — Educational small group session with no FOBT kit
  Other Names: Intervention 2
  Arms: Arm 2
Behavioral: Arm 3 — Educational small group session, exercise
  Other Names: Control
  Arms: Arm 3

SUMMARY:
Develop and evaluate in a randomized trial an educational small group intervention to increase colorectal cancer screening among Filipino Americans.

DETAILED DESCRIPTION:
The purpose of this research study is to increase colorectal cancer (CRC) screening among older Filipino Americans, specifically the use of fecal occult blood tests (FOBTs). We will design a culturally specific intervention, an educational small group discussion with a Filipino health professional. The effect of the intervention will be tested with 620 Filipino Americans. Subjects will be recruited at community-based organizations and churches and invited to join a 1 1/2 hour discussion of health issues with their partner and some of their friends. A third of the subjects will discuss exercise (control group), another third will discuss CRC and receive an FOBT kit, and the remaining third will discuss CRC and will not receive an FOBT kit. Three months after the group session, subjects in the CRC (intervention) groups will receive a letter reminding them to get screened. All subjects will be interviewed before and 6 months after the group sessions to assess CRC screening levels in the three groups. Self-reported CRC screening will be verified by a review of their medical records.

ELIGIBILITY:
Inclusion Criteria:

* Being: a Filipino American,
* Member of or affiliated with participating community agencies, between the ages of 50 and 70,
* Not up-to-date with colorectal cancer screening at baseline

Exclusion Criteria:

* Being younger than 50 or older than 70 years,
* Not being a member or not affiliated with participating community agencies,
* Not being Filipino American or up-to-date with colorectal cancer screening at baseline

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 906 (Actual)
Dates: Start 2004-09; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Receipt of a colorectal cancer screening test | 6 months post-intervention

SECONDARY OUTCOMES:
Knowledge and attitudes regarding CRC screening. | 6 months post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Annette E Maxwell, Dr.P.H., Principal Investigator — University of California, Los Angeles
Locations (1):
- Division of Cancer Prevention and Control Research, Univ of California Los Angeles, Los Angeles, California, United States

REFERENCES:
- [Result] Maxwell AE, Danao LL, Crespi CM, Antonio C, Garcia GM, Bastani R. Disparities in the receipt of fecal occult blood test versus endoscopy among Filipino American immigrants. Cancer Epidemiol Biomarkers Prev. 2008 Aug;17(8):1963-7. doi: 10.1158/1055-9965.EPI-07-2800. PMID 18708385
- [Result] Maxwell AE, Bastani R, Danao LL, Antonio C, Garcia GM, Crespi CM. Results of a community-based randomized trial to increase colorectal cancer screening among Filipino Americans. Am J Public Health. 2010 Nov;100(11):2228-34. doi: 10.2105/AJPH.2009.176230. Epub 2010 Sep 23. PMID 20864724
- [Result] Maxwell AE, Bastani R, Crespi CM, Danao LL, Cayetano RT. Behavioral mediators of colorectal cancer screening in a randomized controlled intervention trial. Prev Med. 2011 Feb;52(2):167-73. doi: 10.1016/j.ypmed.2010.11.007. Epub 2010 Nov 25. PMID 21111754